CLINICAL TRIAL: NCT02192710
Title: Reduction of Preoperative Anxiety in Children: Electronic Tab vs Midazolam
Acronym: IPAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013.794
Record Dates: First submitted 2014-04-25; First posted 2014-07-17 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Paediatric Outpatient Surgery
Keywords: outpatient surgery; anaesthesia; midazolam; electronic tab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnovel® (midazolam) (Active Comparator): Midazolam oral intake before anesthesia
  Interventions: Drug: Midazolam oral intake
- Electronic tab (Experimental)
  Interventions: Procedure: electronic tab

INTERVENTIONS:
Procedure: electronic tab — classic use of an electronic tab with age specific games
  Arms: Electronic tab
Drug: Midazolam oral intake
  Arms: Hypnovel® (midazolam)

SUMMARY:
Rationale:

The most frequently used means to prevent pre-anaesthetic anxiety in children is a drug premedication. Midazolam, a benzodiazepine, is mainly used. It requires time for action, so coordination between departments and operating room, exposed to the risks of side effects and failure and this variability action. Alternative means were evaluated, such as the presence of parents during anaesthetic mask induction, distraction by clowns, hypnosis or video games.

Electronic tabs are small devices; light, easy to use with age-specific and interactive programs. Our hypothesis is that these electronic tabs are more effective in reducing anxiety and distract children compare to preoperative medication.

Methods: This is a monocentric, randomized, open-label study comparing patients aged 4 to 10 years old programmed for a short term and low level of pain outpatient surgery. My pass score will be measured when arriving at the hospital, at the time of the separation with the parents, at the time of the anaesthetic mask induction and after the surgery.

118 patients will be randomized as follows :

* Arm 1 : Hypnovel® (midazolam)
* Arm 2 : Electronic tab The recruitment is performed by general practitioners in the Lyon area.

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys aged 4 to 10 years,
* American Society of Anesthesiologists Score between 1 and 3,
* programmed outpatient surgery for a short term and low level of pain
* Infection with influenza A virus confirmed with a quick diagnostic test,
* informed consent from both parents

Exclusion Criteria:

* patients younger than 4 or older than 10 years old
* preexisting psychiatric disorder with pedo-psychiatric follow-up
* children with intellectual disability
* psychotropic referred to anxiolytic and / or antipsychotic
* history of surgery (n>=3)
* refusal to participate

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Patient's level of anxiety | at day 1
  Comparison of m-YPAS score between the 2 arms at the time of anaesthetic mask induction (H0)

SECONDARY OUTCOMES:
Patient's level of anxiety | At day 1
  Comparison of m-YPAS score between the 2 arms
  * when arriving at the operating room airlock H-1 before surgery,
  * at the time of the separation with the parents
  * 15 minutes before surgery and
  * 30 minutes before departure from the hospital the same day
Parents' level of anxiety | At Day 1
  Evaluation of parents anxiety will be assessed by State-Trait Anxiety Inventory (STAI) :
  * when arriving at the operating room airlock H-1 before surgery,
  * at the time of the separation with the parents
  * 15 minutes before surgery and
  * 30 minutes before departure from the hospital the same day
Parents' level of anxiety | Up to 2 weeks after Day 1
  post-surgery behavioral changes will be measured using the Post Hospitalization Behavioral Questionnaire (PHBQ) at Day+1, day+7 and Day+14 after surgery
Satisfaction of patients, parents and medical team | at day 1
  Evaluation of the general satisfaction of children, parents and anesthetic staff will be measured using Visual Analogic Scale (VAS) 30 minutes before departure from the hospital the same day

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'anesthésie, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Result] Marechal C, Berthiller J, Tosetti S, Cogniat B, Desombres H, Bouvet L, Kassai B, Chassard D, de Queiroz Siqueira M. Children and parental anxiolysis in paediatric ambulatory surgery: a randomized controlled study comparing 0.3 mg kg-1 midazolam to tablet computer based interactive distraction. Br J Anaesth. 2017 Feb;118(2):247-253. doi: 10.1093/bja/aew436. PMID 28100529